CLINICAL TRIAL: NCT05764239
Title: A Phase 3, Double-blind, Placebo-controlled, Randomized Withdrawal Study to Evaluate the Efficacy and Safety of SYNB1934 in Patients With PKU (SYNPHENY-3)
Brief Title: Efficacy and Safety of SYNB1934 in Patients With PKU (SYNPHENY-3)
Acronym: SYNPHENY-3
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Based on a review of interim data from participants in the dose-escalation phase, it was determined that the study was unlikely to meet the primary endpoint.
Sponsor: Synlogic (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SYNB1934-CP-003
Record Dates: First submitted 2023-02-15; First posted 2023-03-10 (Actual); Results first posted 2024-06-20 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-05

CONDITIONS: Phenylketonuria
Keywords: PKU; Inborn error of metabolism; Synpheny; Synlogic; Phe; Metabolic
MeSH Terms: conditions — Phenylketonurias; Metabolism, Inborn Errors

STUDY DESIGN:
Intervention Model Description: This was a Phase 2b/3 adaptive study design.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The DEP (Part 1) and OLE (Part 3) were open label, and the RWP (Part 2) was double blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- DEP (Part 1, SYNB1934v1) (Experimental): Participants received SYNB1934v1 orally immediately after meals on the following dose-ramp regimen:
  Dose level 1 (Days 1-9): 3 × 10^11 live cells partial dose up to 3 times daily (TID); Dose level 2 (Weeks 4-6): 6 × 10^11 live cells up to TID; Dose level 3 (Weeks 7-9): 1 × 10^12 live cells up to TID.
  Interventions: Drug: SYNB1934v1
- RWP (Part 2, SYNB1934v1) (Experimental): Participants who completed the DEP were randomized 1:1 to receive SYNB1934v1 at their iTD established in the DEP orally immediately after meals. Participants remained on this dose of SYNB1934v1 for the duration of the RWP; doses of SYNB1934v1 were not permitted to be modified during the RWP.
  Interventions: Drug: SYNB1934v1
- RWP (Part 2, Placebo) (Placebo Comparator): Participants who completed the DEP were randomized 1:1 to receive placebo orally immediately after meals. Participants remained on the same dose of placebo for the duration of the RWP; doses of placebo were not permitted to be modified during the RWP.
  Interventions: Drug: Placebo
- OLE (Part 3, SYNB1934v1) (Experimental): Participants completed a dose ramp to their iTD guided by tolerability, as described for the DEP, including the full dose-ramp schedule. The iTD in the OLE may have been different from the iTD in the DEP or RWP. The investigator may have escalated the dose of SYNB1934v1 up to 1 × 10^12 live cells based on tolerability; multiple attempts to escalate to a higher dose level were permitted per investigator discretion.
  Interventions: Drug: SYNB1934v1

INTERVENTIONS:
Drug: SYNB1934v1 — SYNB1934v1 consisted of powder for oral suspension packaged in sachets. During dose preparation, the powder was resuspended in water or apple juice prior to administration.
  Arms: DEP (Part 1, SYNB1934v1); OLE (Part 3, SYNB1934v1); RWP (Part 2, SYNB1934v1)
Drug: Placebo — Placebo was manufactured using an inactive powder that was color matched to the SYNB1934v1 drug product. In order to maintain study blinding during the RWP, placebo was packaged, labeled, stored, and administered in an identical manner to SYNB1934v1.
  Arms: RWP (Part 2, Placebo)

SUMMARY:
SYNB1934-CP-003 was designed as a 3-part, adaptive study consisting of a dose-escalating, open-label period (DEP; Part 1) of up to 15 weeks, followed by a 4-week, double-blind, placebo-controlled, randomized withdrawal period (RWP; Part 2), and an open-label extension (OLE; Part 3) of up to 36 months

DETAILED DESCRIPTION:
In the DEP, all enrolled participants maintained a stable diet reflecting their baseline phenylalanine (Phe) intake and received escalating doses of SYNB1934v1 from approximately 3 to 15 weeks to determine an individually titrated dose (iTD), which was defined as the highest dose the participant was able to tolerate. A participant was defined as having reached an iTD if they tolerated 3 weeks at a dose, regardless of whether other doses were tolerated.

Blood Phe level was measured at each dose level after 3 weeks at that level. A responder was defined as a participant who achieved a ≥ 20% reduction in blood Phe level compared to DEP baseline on SYNB1934v1.

Participants who completed at least 3 weeks at their iTD during the DEP entered a 4-week RWP in which they were randomized 1:1 to receive SYNB1934v1 at their iTD determined in the DEP or placebo TID. Randomization was stratified on screening Phe level. Participants remained on their assigned dose (iTD of SYNB1934v1 or matching placebo) for the duration of the RWP, unless they developed intolerance or met other discontinuation criteria, and remained on the same diet they consumed during the DEP. Blood Phe level was measured at Weeks 1, 3, and 4 of the RWP.

Participants who completed the 4-week RWP may have entered the OLE and received SYNB1934v1 for up to 36 months. During the OLE, participants completed a dose ramp to their iTD over time guided by tolerability. The iTD in the OLE may have been different from the iTD in the DEP. The investigator may have escalated the SYNB1934v1 dose up to 1 × 10^12 live cells based on tolerability. Participants were allowed to modify their standard diet, with guidance from the investigator, if their blood Phe level was < 240 µmol/L.

ELIGIBILITY:
Male and female participants were enrolled.

Inclusion Criteria:

1. Age ≥ 18 years.
2. Able and willing to voluntarily complete the informed consent process.
3. Diagnosis of phenylketonuria (PKU) and failure to maintain recommended blood Phe levels on existing management (sapropterin, sepiapterin, and/or Phe-restricted diet), demonstrated by uncontrolled blood Phe level > 360 μmol/L on current therapy any time during screening and uncontrolled blood Phe level > 360 μmol/L on current therapy when taking the average of the 3 most recent Phe levels from the participant's medical history (inclusive of any screening values). All screening values must have been obtained more than 7 days apart, as determined by central or local laboratory.
4. Females of childbearing potential must have had a negative pregnancy test at screening and at the end of the DEP (in order to enter the RWP) and RWP (in order to enter the OLE) and been willing to have additional pregnancy tests during the study.
5. Sexually active female participants of childbearing potential must have been willing to use an acceptable method of contraception while participating in the study and for 2 weeks after the last dose.
6. Stable diet including stable medical formula regimen (if used) for at least 1 month prior to screening.
7. If using sapropterin or sepiapterin, must have been on a stable dose for at least 3 months.
8. Willing and able to continue current diet, sapropterin, sepiapterin, and large neutral amino acids unchanged during screening, DEP, and RWP and to engage in all study activities.

Exclusion Criteria:

1. Currently taking Palynziq® (pegvaliase-pqpz) (within 1 month of screening).
2. Acute or chronic medical, surgical, psychiatric, or social condition or laboratory abnormality that may have increased participant risk associated with study participation, compromised adherence to study procedures and requirements, and, in the judgment of the investigator, would have made the participant inappropriate for enrollment.
3. A known or suspected diagnosis of DNAJC12 deficiency, biopterin synthesis deficiency, or irritable bowel syndrome.
4. Intolerance to or allergic reaction to Escherichia coli Nissle or any of the ingredients in SYNB1934v1 formulation, or an allergy to cinnamon. Known intolerance to proton pump inhibitors and H2 blockers, since one or the other must have been used.
5. Currently taking or plans to take any type of systemic (e.g., oral or intravenous) antibiotic within 28 days prior to the first dose of SYNB1934v1 through final safety assessment in the RWP, including planned surgery, hospitalizations, dental procedures, or interventional studies that were expected to require antibiotics. Exception: topical antibiotics were allowed.
6. Pregnant, planning to become pregnant, or breastfeeding.
7. Current participation in any other investigational drug study or use of any investigational agent within 30 days or 5 half-lives (whichever was longer) prior to screening.
8. Ever received gene therapy for treatment of PKU.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2023-07-05 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2024-03-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (21):
- United States (14):
  - Science 37, Culver City, California
  - Children's Hospital Orange County, Orange, California
  - Stanford University, Department of Pediatrics, Palo Alto, California
  - University of Colorado Children's Hospital, Aurora, Colorado
  - University of Florida - Gainesville, Gainesville, Florida
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Pediatrics, Chicago, Illinois
  - Massachusetts General Hospital, Department of Pediatrics, Boston, Massachusetts
  - Oregon Health and Science University Department of Molecular and Medical Genetics, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Pediatrics, Charleston, South Carolina
  - Division of Medical Genetics-Pediatrics, Vanderbilt University Medical Center, Nashville, Tennessee
  - UT Southwestern Medical Center, Dallas, Texas
  - McGovern Medical School/Memorial Hermann Hospital, Houston, Texas
- Canada (4):
  - MAGIC Clinic, Calgary, Alberta
  - Hamilton Health Sciences Corporation, Hamilton, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - University Health Network, Toronto, Ontario
- Medical Genetics and Laboratory Diagnostics Center, Tbilisi, Georgia
- Turkey (Türkiye) (2):
  - Gazi Üniversitesi Hastanesi, Yenimahalle, Ankara
  - Dokuz Eylül Üniversitesi Araştırma ve Uygulama Hastanesi, Balçova, İzmir

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- All Participants: In the DEP (Part 1), participants received SYNB1934v1 on the following dose-ramp regimen:
  Dose level 1 (Days 1-9): 3 × 10^11 live cells partial dose up to TID; Dose level 2 (Weeks 4-6): 6 × 10^11 live cells up to TID; Dose level 3 (Weeks 7-9): 1 × 10^12 live cells up to TID.
  In the RWP (Part 2), participants who completed the DEP were randomized 1:1 to receive SYNB1934v1 at their iTD established in the DEP (no modifications permitted).
  In the OLE (Part 3), participants completed a dose ramp to their iTD guided by tolerability, as described for the DEP, including the full dose-ramp schedule; the OLE iTD may have been different from the DEP/RWP iTD.
  SYNB1934v1 and placebo (color matched) consisted of powder for oral suspension packaged in sachets and resuspended in water or apple juice. Investigational medical product (IMP, ie, SYNB1934v1 or placebo) was administered orally immediately after meals.
Period: DEP (Part 1)
Arm/Group | All Participants
Started | 35
Completed DEP | 17
Completed (Completed study) | 0
Not Completed | 35
Not completed — Study terminated by Sponsor | 28
Not completed — Withdrawal by Subject | 3
Not completed — Non-compliance with study drug | 2
Not completed — Adverse Event | 1
Not completed — Lost to Follow-up | 1
Period: RWP (Part 2, SYNB1934v1)
Arm/Group | All Participants
Started | 9
Completed RWP | 9
Completed (Completed study) | 0
Not Completed | 9
Not completed — Study terminated by Sponsor | 7
Not completed — Non-compliance with study drug | 2
Period: RWP (Part 2, Placebo)
Arm/Group | All Participants
Started | 8
Completed RWP | 8
Completed (Completed Study) | 0
Not Completed | 8
Not completed — Study terminated by Sponsor | 8
Period: OLE (Part 3)
Arm/Group | All Participants
Started | 10
Completed (Completed OLE and/or study) | 0
Not Completed | 10
Not completed — Study terminated by Sponsor | 10

BASELINE CHARACTERISTICS:
Population: All participants who took at least 1 dose of SYNB1934v1 in the indicated study period (DEP or OLE) or who were randomized into the RWP.
Groups:
- All Participants: In the DEP (Part 1), participants received SYNB1934v1 on the following dose-ramp regimen:
  Dose level 1 (Days 1-9): 3 × 10^11 live cells partial dose up to TID; Dose level 2 (Weeks 4-6): 6 × 10^11 live cells up to TID; Dose level 3 (Weeks 7-9): 1 × 10^12 live cells up to TID. In the RWP (Part 2), participants who completed the DEP were randomized 1:1 to receive SYNB1934v1 at their iTD established in the DEP (no modifications permitted).
  In the OLE (Part 3), participants completed a dose ramp to their iTD guided by tolerability, as described for the DEP, including the full dose-ramp schedule; the OLE iTD may have been different from the DEP/RWP iTD.
  SYNB1934v1 and placebo (color matched) consisted of powder for oral suspension packaged in sachets and resuspended in water or apple juice. IMP was administered orally immediately after meals.
Arm/Group | All Participants
Number analyzed (Participants) | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 35
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: years] | 31.0 [18 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 33
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 30
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  Canada | 10
  United States | 25

OUTCOME MEASURES:

1. Primary Outcome: Mean Percent Change From DEP Baseline in Blood Phenylalanine (Phe) Level at Week 3 of iTD During the DEP
Description: Baseline for blood Phe level in the DEP was defined as the mean of the duplicate blood Phe level measurements obtained immediately prior to administration of the first dose in the DEP. If only 1 blood Phe level measurement was available, then that measure was used as baseline. The last measurement was the participant's last Week 3 blood Phe level at the iTD of SYNB1934v1.
Time Frame: Up to 15 weeks
Population: Participants who received at least 1 dose of IMP during the DEP, achieved an iTD, and had Week 3 blood Phe measured.
Measure: Median (Full Range); unit: percent change
Groups:
- iTD of 3 x 10^11 Live Cells; iTD of 6 x 10^11 Live Cells; iTD of 1 x 10^12 Live Cells; Overall DEP: Participants received SYNB1934v1 orally immediately after meals.
  SYNB1934v1 consisted of powder for oral suspension packaged in sachets and resuspended in water or apple juice prior to administration.
Arm/Group | iTD of 3 x 10^11 Live Cells | iTD of 6 x 10^11 Live Cells | iTD of 1 x 10^12 Live Cells | Overall DEP
Number analyzed (Participants) | 0 | 1 | 14 | 15
percent change |  | -3.85 [0 to -3.85] | 5.33 [-37.2 to 59.3] | 3.35 [-37.2 to 59.3]

2. Secondary Outcome: Absolute Change From DEP Baseline in Blood Phe Level at Week 3 of iTD During the DEP
Description: as for outcome 1
Time Frame: Up to 15 weeks
Population: Participants who received at least 1 dose of IMP during the DEP, achieved an iTD, and had Week 3 blood Phe measured.
Measure: Median (Full Range); unit: µmol/L
Arm/Group | iTD of 3 x 10^11 Live Cells | iTD of 6 x 10^11 Live Cells | iTD of 1 x 10^12 Live Cells | Overall DEP
Number analyzed (Participants) | 0 | 1 | 14 | 15
µmol/L |  | -55.00 [0 to -55.00] | 55.25 [-227.0 to 406.5] | 30.50 [-227.0 to 406.5]

3. Secondary Outcome: Number of Participants With a ≥ 20% Reduction From Baseline in Blood Phe Level at Any Time in the DEP
Description: Baseline for blood Phe level in the DEP was defined as the mean of the duplicate blood Phe level measurements obtained immediately prior to administration of the first dose in the DEP. If only 1 blood Phe level measurement was available, then that measure was used as baseline. Blood Phe level was measured at each dose level after 3 weeks at that level.
Time Frame: Up to 15 weeks
Population: Participants who received at least 1 dose of IMP during the DEP, achieved an iTD, and had blood Phe measured.
Measure: Count of Participants; unit: Participants
Arm/Group | iTD of 3 x 10^11 Live Cells | iTD of 6 x 10^11 Live Cells | iTD of 1 x 10^12 Live Cells | Overall DEP
Number analyzed (Participants) | 1 | 1 | 15 | 17
Participants | 0 | 0 | 6 | 6

ADVERSE EVENTS:
Time Frame: All AEs occurring from the time a participant signed the informed consent form through the safety follow-up period and at least 1 month following the last dose of IMP were documented, regardless of causal assessment to IMP.
Description: Adverse event (AE) documentation included duration (start and end dates or ongoing), severity using the Common Terminology Criteria for Adverse Events (version 5.0), assessment of causality, and whether specific action or therapy was required. Within each study period, each AE term is counted only once per participant at the maximum reported grade.
Groups:
- DEP (Part 1, SYNB1934v1): Participants received SYNB1934v1 orally immediately after meals on the following dose-ramp regimen:
  Dose level 1 (Days 1-9): 3 × 10^11 live cells partial dose up to TID; Dose level 2 (Weeks 4-6): 6 × 10^11 live cells up to TID; Dose level 3 (Weeks 7-9): 1 × 10^12 live cells up to TID.
  SYNB1934v1 consisted of powder for oral suspension packaged in sachets and resuspended in water or apple juice prior to administration.
- RWP (Part 2, SYNB1934v1): Participants who completed the DEP were randomized 1:1 to receive SYNB1934v1 at their iTD established in the DEP orally immediately after meals. Participants remained on this dose of SYNB1934v1 for the duration of the RWP.
  SYNB1934v1 consisted of powder for oral suspension packaged in sachets and resuspended in water or apple juice prior to administration.
- RWP (Part 2, Placebo): Participants who completed the DEP were randomized 1:1 to receive placebo orally immediately after meals. Participants remained on this dose of placebo for the duration of the RWP.
  Placebo consisted of inactive powder (color matched to SYNB1934v1) for oral suspension packaged in sachets and resuspended in water or apple juice prior to administration.
- OLE (Part 3, SYNB1934v1): Participants completed a dose ramp to their iTD guided by tolerability, as described for the DEP, including the full dose-ramp schedule. The iTD in OLE may have been different from the iTD in the DEP or RWP.
  SYNB1934v1 consisted of powder for oral suspension packaged in sachets and resuspended in water or apple juice prior to administration.
Arm/Group | DEP (Part 1, SYNB1934v1) | RWP (Part 2, SYNB1934v1) | RWP (Part 2, Placebo) | OLE (Part 3, SYNB1934v1)
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/9 | 0/8 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/9 | 0/8 | 0/10
Other Adverse Events (participants affected / at risk) | 23/35 | 3/9 | 5/8 | 2/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DEP (Part 1, SYNB1934v1) (N=35) | RWP (Part 2, SYNB1934v1) (N=9) | RWP (Part 2, Placebo) (N=8) | OLE (Part 3, SYNB1934v1) (N=10)
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 11 | 0 | 0 | 1
Flatulence (Gastrointestinal disorders) | 9 | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 7 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 7 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 5 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 5 | 0 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Faeces soft (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastrointestinal sounds abnormal (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Fatigue (General disorders) | 2 | 0 | 0 | 0
Influenza like illness (General disorders) | 1 | 2 | 1 | 0
Nasopharyngitis (Infections and infestations) | 5 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 3 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 1 | 0
Oral herpes (Infections and infestations) | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Wound infection (Infections and infestations) | 1 | 0 | 0 | 0
Weight decreased (Investigations) | 1 | 0 | 0 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Subchondral insufficiency fracture (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 3 | 0 | 0 | 2
Sinus headache (Nervous system disorders) | 1 | 0 | 0 | 0
Affect lability (Psychiatric disorders) | 1 | 0 | 0 | 0
Agitation (Psychiatric disorders) | 1 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 0
Mood swings (Psychiatric disorders) | 1 | 0 | 0 | 0
Ovarian cyst (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Viral infection (Infections and infestations) | 0 | 0 | 1 | 0
Eye infection (Infections and infestations) | 0 | 1 | 0 | 0
Folliculitis (Infections and infestations) | 0 | 1 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Memory impairment (Nervous system disorders) | 0 | 0 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of participants analyzed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2023-07-01): https://cdn.clinicaltrials.gov/large-docs/39/NCT05764239/Prot_000.pdf
  • Statistical Analysis Plan (2023-10-05): https://cdn.clinicaltrials.gov/large-docs/39/NCT05764239/SAP_001.pdf